CLINICAL TRIAL: NCT05438992
Title: Comparing the Effect of Three Different Volumes of Bupivacaine in Infiltration Between Popliteal Artery and Capsule of Knee Block Following Adductor Canal Block in Total Knee Arthroplasty, Prospective Randomized Control Trial.
Brief Title: Different Bupivacaine Volumes in Infiltration Between Popliteal Artery and Capsule of Knee Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Omar Ahmed, Associate professor of Anesthesia, pain management & surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-339-2021
Record Dates: First submitted 2022-06-25; First posted 2022-06-30 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): The patients in this group will be administered 15 ml bupivacaine 0.250 % between the popliteal artery and the capsule of the posterior knee.
  Interventions: Drug: Bupivacaine 0.25% Preservative-Free Injectable Solution
- Group B (Active Comparator): The patients in this group will be administered 20 ml bupivacaine 0.250 % between the popliteal artery and the capsule of the posterior knee.
  Interventions: Drug: Bupivacaine 0.25% Preservative-Free Injectable Solution
- Group C (Active Comparator): The patients in this group will be administered 25 ml bupivacaine 0.250 % between the popliteal artery and the capsule of the posterior knee.
  Interventions: Drug: Bupivacaine 0.25% Preservative-Free Injectable Solution

INTERVENTIONS:
Drug: Bupivacaine 0.25% Preservative-Free Injectable Solution — local anesthetic drug injection for postoperative pain

SUMMARY:
comparing between three different volumes; 15, 20 & 25 ml of 0.25% bupivacaine to determine the best volume of Infiltration Between Popliteal Artery and Capsule of Knee (IPACK) block following adductor canal block (ACB) with the best analgesia and least complications after total knee arthroplasty (TKA)

DETAILED DESCRIPTION:
105 participants will be randomized into three groups based on computer generated numbers using online randomization program

Preoperative assessment is conducted on the patients that will be enrolled in this study including history taking, physical examination, and routine laboratory investigations; in the form of CBC, coagulation profile, creatinine, urea, ALT, AST and radiological investigations; according to the medical condition of the patients. All patients should fulfill the inclusion criteria.

a written informed consent form will be obtained from the patients that will be enrolled in the study.

Preoperative:

On the day of surgery, the patient ID will be confirmed in the preparation room, then 18 G cannula will be inserted to the patient, premedication will be given including lactated ringer solution 500 ml, midazolam 2 mg & metoclopramide 10 mg.

VAS scale. Visual analogue scale (VAS) for measuring post-operative pain will be explained to all patients. VAS is a horizontal line, 100 mm in length, anchored by word descriptors at each end. It has two ends one end was labelled as no pain (0) and the other end was labelled as worst pain (10)".

The patient marks on the line the point that they feel represents their perception of their current state.

Intraoperative:

The patients enrolled in the study will be transferred to the Operation room and monitored all through the surgical procedure using pulse oximeter, non-invasive blood pressure and ECG.

To perform spinal anesthesia ,the patient will be positioned in the sitting position then sterilization of the back using betadine solution 5% will be done then the iliac crest will be identified and the opposite intervertebral space(L4-L5) will be marked then 5 ml of lidocaine 2% will be infiltrated in the skin and subcutaneous tissue then a spinal needle (22 G )or(25 G) will be introduced to the intrathecal space and after ensuring that clear cerebrospinal fluid will be in free flow injection of 15 - 20 mg of bupivacaine 0.5 % and 25 mcg of fentanyl will be administrated then the patient will be positioned in the supine position.

If hypotension, (decrease in the mean arterial blood pressure of more than 20%from base line) occurs, 3mg ephedrine will be given with 200ml bolus crystalloids. If bradycardia (heart rate below 50 beat / minute) occurs, 0.5 mg intravenous atropine will be given.

At the end of the operation, patients will be randomly allocated using computerized generated random tables in to three equal groups and the random numbers will be concealed in closed opaque envelopes which will be kept by the senior anesthesia staff, the three groups are:

Group A: The patients in this group will be administered 15 ml bupivacaine 0.250 % between the popliteal artery and the capsule of the posterior knee.

Group B: The patients in this group will be administered 20 ml bupivacaine 0.250 % between the popliteal artery and the capsule of the posterior knee.

Group C: The patients in this group will be administered 25 ml bupivacaine 0.250 % between the popliteal artery and the capsule of the posterior knee.

With the patient in the supine position, adductor canal block will be performed, the procedural needle will be inserted in-plane from the anteromedial side at the mid-thigh level. It will be advanced through the sartorius muscle and fascia under ultrasound guidance, using a Siemens Acuson X300 ultrasound equipped with a linear transducer after sterilization of the skin with betadine solution 5%, and the adductor canal, with the superficial femoral artery and vein within, will be identified. Once the needle ( spinal needle 22g) tip will be located in the adductor canal, 20 ml bupivacaine 0.25% will be injected anterior to the artery and deep into the sartorius muscle.

.

Then, IPACK block will be performed by scanning the popliteal fossa under ultrasound guidance, the transducer will be slowly moved toward the popliteal crease until the tibial nerve will be identified superficial to the popliteal vessels. The femoral condyles will be defined at this level. The needle will be advanced in a medial- to- lateral direction using an in plane approach and advanced to the intercondylar fossa between the popliteal artery and the femoral condyles. When the needle tip will be located anteriorly to the lateral edge of the popliteal artery, the volume of bupivacaine 0.250% according to each group will be injected using spinal needle 22 gauge while slowly withdrawing the needle until the tip of the needle reached the medial femoral condyle. After that patient will be transferred to the recovery room then to the ward.

Patient should be will monitored during injection of local anesthetic to detect local anesthetic toxicity which usually begins within 1-5 min and may delay up to 1 hr with prodromal signs, as perioral numbness, tinnitus, agitation, dysarthria, and confusion. Then severe central nervous system (CNS) symptoms such as seizures and coma. Also, cardiovascular( CV) symptoms presenting initially with hypertension and tachycardia, then bradycardia and hypotension, with progression to more serious complications, including ventricular arrhythmias and asystole. The patient can manifest as isolated CV dysfunction or as a combination of CNS and CV signs without the classical progression.

Risk of toxicity increases with the type of local anesthetic and dose, site of injection, extremes of age and patient's comorbidities as organ dysfunction, Preexisting cardiac disease which increase risk of arrhythmias and myocardial depression and the serum level of the binding proteins.

So caution is advised in patient with decompensated heart failure, severe valvular disease, or depressed ventricular function. Also, Patients with renal or hepatic failure can result in decreased metabolism and clearance and a higher level of circulating drug. In addition, malnutrition, or any other disease process that results in a decreased serum level of albumin can increase the level of the free drug for a given dose.

Postoperative:

1. Postoperative pain will be assessed by visual analog scale (VAS) at times 0-30 minutes, 1, 2, 4, , 8, 12, 18 and 24 hours postoperatively.
2. Postoperative pain assessment through VAS will be according to the scale as follow:

   * Pain level 0: no pain
   * Pain level1-3: mild pain
   * Pain level 4-6: moderate pain
   * Pain level 7-10: severe pain
3. Postoperative pain will be managed as follow:

   * Mild pain will be treated with paracetamol 1 gm iv.
   * Moderate pain will be treated with paracetamol 1 gm iv & ketolac, 30 mg iv.
   * Severe pain will be treated with paracetamol 1 gm iv , ketolac, 30 mg iv & morphine 0.1 mg/kg iv (rescue analgesia) Then patient will be reassessed and recorded as mentioned above and the specific treatment will be repeated after 8 hours from the initial dose according to VAS.
4. Opioids complications such as respiratory depression will be recorded and managed supportively by oxygen mask, controlled airway and if persistent or severe hypoventilation occurs positive pressure ventilation may be needed, nausea and vomiting will be treated with ondansetron (4 mg IV).
5. Criteria of failed block : persistent sever pain after elimination of spinal anesthesia vas score >6 and need more doses of opioids

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing knee arthroscopy surgery.
* Age between 18 years and 65 years.
* Both sexes
* ASA I & ASA II

Exclusion Criteria:

* Patients' refusal
* Allergy to any drug that will be used in the study
* Psychological or mental disorders.
* Disturbance of Conscious level.
* Uncooperative patients
* Coagulopathy
* Contraindications to spinal anaesthesia (e.g.: severe mitral stenosis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
visual analogue score ( VAS) for 24 hours postoperatively | 24 hours
  assessment of pain score

SECONDARY OUTCOMES:
first rescue analgesia time | 24 hours
  Time (in hours) of first rescue analgesia (morphine 0.1mg/kg) requirement for each group following the IPACK block
morphine consumption | 24 hours
  Total amount of morphine/kg consumed in the first 24 hours following the IPACK block ( Max dose 0.4mg/kg/24hrs).
sensory block | 24 hours
  duration of sensory block through 24hrs using test ice.
morphine complications | 24 hours
  nausea and vomiting, bradycardia, respiratory depression
postoperative hemodynamics | 24 hours
  postoperative hemodynamics including heart rate, blood pressure at times 0-30 minutes, 1, 2, 4, , 8, 12, 18 and 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Heba Omar, MD, Principal Investigator — associate professor of anesthesia and surgical ICU, faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No